CLINICAL TRIAL: NCT02417688
Title: PET-MR Imaging of Natriuretic Peptide Receptor C (NPR-C) in Carotid Atherosclerosis With [64]Cu-25%CANF-Comb
Brief Title: PET Imaging of Natriuretic Peptide Receptor C (NPR-C) in Carotid Atherosclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201409006
Record Dates: First submitted 2015-04-11; First posted 2015-04-16 (Estimated); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Carotid Atherosclerosis
Keywords: carotid atherosclerosis, PET imaging agent
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cu[64]-25%-CANF-Comb PET-MR (Experimental): Single IV injection of 4-8 mCi of Cu[64]-25%-CANF-Comb with a mass no more than 100 μgrams followed by PET-MR Imaging
  Interventions: Device: Cu[64]-25%-CANF-Comb PET-MR

INTERVENTIONS:
Device: Cu[64]-25%-CANF-Comb PET-MR — Single IV injection of a novel radiopharmaceutical for diagnostic imaging of atherosclerosis by PET-MR
  Other Names: Cu[64]-25%-CANF-Comb

SUMMARY:
To demonstrate feasibility of imaging Cu[64]-25%-CANF-Comb uptake in the atherosclerosis of the carotid artery of patients for whom carotid artery endarterectomy surgery is planned in comparison to the carotid artery for which intervention is not planned.

DETAILED DESCRIPTION:
This study is a single center, open-label baseline controlled imaging study designed to demonstrate feasibility of PET imaging of radiopharmaceutical nanoparticle Cu[64]-25%CANF-Comb uptake by PET-MR. Patients will undergo Cu[64]-25%CANF-Comb PET-MR imaging of both carotid arteries. Both carotid arteries will be imaged at the same time. We hope to demonstrate differences in PET SUV (Standardized Uptake Value) in the significantly atherosclerotic artery in patients who will be going to carotid endarterectomy surgery in comparison to the PET SUV in the artery that is not significantly diseased (ie; the artery that will not undergo surgery) . We also will determine whether PET SUV of the Cu[64]-25%CANF-Comb by the plaque correlates to the American Heart Association classifications of atherosclerosis and tissue presence of NPR-C in the ex vivo carotid endarterectomy specimen post surgery as measured by RT-PCR.

ELIGIBILITY:
Inclusion Criteria:

* Patients with carotid atherosclerosis
* Patients must be scheduled for carotid intervention (endarterectomy surgery)
* Signed informed consent.

Exclusion Criteria:

* Unstable clinical conditions
* Pregnancy and lactation
* Inability to lie still for up to 60 min with arms down at sides for PET-MR imaging
* Unwilling to comply with study procedures and unavailable for the duration of the study.
* Pacemakers, brain aneurysm clip, shrapnel and other typical contraindications for MRI imaging.
* Inability to provide written informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-04-05 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
PET SUV (Standardized Uptake Value) | 22-26 hours
  Difference in SUV between the carotid with atherosclerosis (carotid artery to be undergo surgery) and the carotid artery without significant disease (artery for which surgery is not planned).

CONTACTS AND LOCATIONS:
Overall Officials: Pamela K Wooderd, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St.Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators may share your images with other researchers. They may be doing research in areas similar to this research or in other unrelated areas. These researchers may be at Washington University, at other research centers and institutions, or industry sponsors of research. The investigators may also share your research data with large data repositories (a repository is a database of information) for broad sharing with the research community. If the individual research data is placed in one of these repositories only qualified researchers, who have received prior approval from individuals that monitor the use of the data, will be able to look at the information.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Beginning 3 months and ending 10 years following article publication.
Access Criteria: Proposals should be directly submitted to pwoodard@wustl.edu.

REFERENCES:
- [Background] Liu Y, Pressly ED, Abendschein DR, Hawker CJ, Woodard GE, Woodard PK, Welch MJ. Targeting angiogenesis using a C-type atrial natriuretic factor-conjugated nanoprobe and PET. J Nucl Med. 2011 Dec;52(12):1956-63. doi: 10.2967/jnumed.111.089581. Epub 2011 Nov 2. PMID 22049461
- [Background] Liu Y, Abendschein D, Woodard GE, Rossin R, McCommis K, Zheng J, Welch MJ, Woodard PK. Molecular imaging of atherosclerotic plaque with (64)Cu-labeled natriuretic peptide and PET. J Nucl Med. 2010 Jan;51(1):85-91. doi: 10.2967/jnumed.109.066977. Epub 2009 Dec 15. PMID 20008978